CLINICAL TRIAL: NCT04855097
Title: Evaluation of Blood Volume Analysis- Guided Management of Decompensated Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daxor Corporation (Industry)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVA for inpatient HF
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart Failure; Blood Volume
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, two-center, parallel design, interventional, single-blinded pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and treating physicians will have no access to the BVA data in the Standard Care arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard care group (Experimental): Blood Volume Analysis will be performed at admission, during inpatient stay if warranted, and prior to hospital discharge. Treating physicians will be blinded to the results and will choose between a low-moderate and high diuretic dose based on usual care clinical assessment of volume status.
  Interventions: Diagnostic Test: BVA-100
- BVA-guided treatment arm (Experimental): Blood Volume Analysis will be performed at admission, during inpatient stay if warranted, and prior to hospital discharge. Treating physicians will receive the results and will choose between a low-moderate and high diuretic dose based on measured volume status.
  Interventions: Diagnostic Test: BVA-100

INTERVENTIONS:
Diagnostic Test: BVA-100 — The BVA-100 is a medical device that calculates human blood volume using the method of tracer dilution. The device utilizes a tracer of human serum albumin tagged with iodine-131 to measure injected intravascularly and a series of timed blood draws. The amount of tracer in each blood draw is used to calculate the unknown blood volume. Data inputs come from the measured characteristics of subject blood samples (hematocrit and tracer concentration) and tracer calibration standards. The package also calculates the subject expected (or ideal) blood volume from physical parameters. Hyper- or hypovolemia, associated red blood cell volumes, and tracer transudation rate are reported, with statistics showing the quality of the results.

SUMMARY:
Diuretic therapy is first-line treatment for acute decompensated heart failure. However, accurate assessment and management of patient blood volume is challenged by the limitations of physical exam and surrogate markers for blood volume. The study primary objective is to determine if goal-directed care as quantified by direct Blood Volume Analysis (Daxor BVA-100™) in addition to usual care results in more appropriate treatment and consistent achievement of euvolemia.

DETAILED DESCRIPTION:
Over 6 million Americans suffer from heart failure, one of the most prevalent and deadly diseases in the United States. High rates of rehospitalization and mortality and treatment costs have persisted for decades despite advances in care. Clinical guidelines recommend assessment of blood volume and clinical management to euvolemia or normal blood volume, but standard methods of diagnosing blood volume status have been shown to be unreliable. Blood Volume Analysis (Daxor BVA-100) is based on the gold standard indicator dilution technique. BVA has been used to quantify otherwise undiagnosed blood volume derangements and guide treatment in heart failure and other indications. Also, retrospective analyses have shown that care of heart failure patients guided by BVA is associated with improved rates of rehospitalization and mortality.

The proposed study is a prospective, two-center, parallel design, interventional, single-blinded pilot study of the potential for BVA to positively impact the treatment decisions of ADHF clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years. In accordance with the Inclusion Across the Lifespan policy, Children will be excluded from the proposed study. ADHF is a condition that rarely affects children and Daxor's BVA-100 lack the reference norms for pediatric use.
2. Admission to the hospital with a primary diagnosis of ADHF.
3. Able and willing to provide informed written consent.

Exclusion Criteria:

1. Evidence of acute coronary syndrome or myocardial infarction during qualifying ADHF hospitalization.
2. Evidence of hypertensive crisis or acute valvular regurgitation.
3. The following has occurred within the last 3 months or is planned within the following 3 months:

   1. Revascularization procedure.
   2. Placement on cardiac transplantation list.
   3. Other major cardiac surgery or other surgery.
4. Planned intermittent or continuous intravenous positive inotropic therapy.
5. Severe chronic kidney disease (eGFR<15 ml/min).
6. Psycho-social factors that interfere with ability to adhere to study procedures (severe dementia, active substance abuse, poorly controlled psychiatric illnesses).
7. Pregnant women or nursing mothers.
8. Women of childbearing potential not using adequate birth control methods.
9. Known hypersensitivity to iodine or eggs.
10. Participation in another heart failure investigational treatment protocol currently or <30 days prior to enrollment.
11. Evidence of active bleeding or active hemolysis.
12. Hemoglobin measured below 7 g/dl or hematocrit measured below 21%.
13. Patient has received a heart transplant and/or currently treated with mechanical circulatory support.
14. Patients implanted with invasive hemodynamic monitors (i.e. CardioMEMS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Quantitative assessment of progress to euvolemic target for both subjects and controls | Approximately 2 weeks
  Accurately quantify levels and changes to blood volume and red blood cell volume in ADHF inpatients during inpatient stay, and use this data to guide diuretic therapy in the treatment arm.

SECONDARY OUTCOMES:
Quantitative assessment of event-based outcome metrics | 30 days post discharge
  30-day readmission and mortality outcomes will be quantified for both cohorts.
Quantitative assessment of continuous outcome metrics: weight | Approximately 2 weeks
  Measure and compare changes to body weight in kilogram
Quantitative assessment of continuous outcome metrics: net fluid balance | Approximately 2 weeks
  Measure and compare changes to net fluid balance in mL
Quantitative assessment of continuous outcome metrics: natriuretic peptide | Approximately 2 weeks
  Measure and compare changes to natriuretic peptide in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Joseph, Principal Investigator — Boston VA Healthcare System; Bradley Bart, Principal Investigator — Minneapolis Veterans Affairs Medical Center; Orly Vardeny, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will primarily be captured from Clinical Report Forms and de-identified data will be transferred from the clinical sites to Daxor for analysis. All PHI used to abstract data will remain on the VA Health System servers and will not be transported outside for any research purpose. In accordance with VA policy, incident reporting of theft, loss of data, loss of storage media, unauthorized access to sensitive data or storage media and non-compliance with security controls will be reported promptly to the study PI, Privacy Officer and Information Security Officer.
Supporting Information: CSR
Time Frame: Data will become available as collected throughout the study, and will be available for 18months prior to the completion of the study, for analysis.